CLINICAL TRIAL: NCT01065636
Title: Exercise Interventions During Voluntary Weight Loss in Obese Older Adults
Brief Title: Lifestyle Intervention Trial in Obese Elderly
Acronym: LITOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomedical Research Institute of New Mexico (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Dennis Villareal, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AG031176 (NIH); R01AG031176 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diet + Resistance Exercise Training (Experimental): Weekly behavioral/diet-induced weight loss plus supervised resistance exercise training three times a week
  Interventions: Behavioral: Diet + Resistance Training
- Diet + Aerobic Exercise Training (Experimental): Weekly behavioral/diet-induced weight loss plus supervised aerobic exercise training three times a week
  Interventions: Behavioral: Diet + Aerobic Training
- Diet + Combined Aerobic/Resistance Exercise (Experimental): Weekly behavioral/diet-induced weight loss plus combined supervised resistance exercise training and aerobic exercise training three times a week
  Interventions: Behavioral: Diet + Resistance/Aerobic Exercise
- Control Group (No Diet/No Exercise) (No Intervention): No diet No exercise training

INTERVENTIONS:
Behavioral: Diet + Resistance Training — Behavioral Therapy through a lifestyle modification program, Diet therapy once weekly through a dietician prescribed diet for 26 weeks, and resistance exercise training 3-days/week for 24 weeks.
  Arms: Diet + Resistance Exercise Training
Behavioral: Diet + Aerobic Training — Behavioral Therapy through a lifestyle modification program, Diet therapy once weekly through a dietician prescribed diet for 26 weeks, and aerobic exercise training 3-days/week for 24 weeks
  Arms: Diet + Aerobic Exercise Training
Behavioral: Diet + Resistance/Aerobic Exercise — Behavioral Therapy through a lifestyle modification program, Diet therapy once weekly through a dietician prescribed diet for 26 weeks, and combined resistance/aerobic exercise training 3-days/week for 24 weeks
  Arms: Diet + Combined Aerobic/Resistance Exercise

SUMMARY:
Obesity causes frailty in obese older adults by exacerbating the age-related decline in physical function. However, appropriate management of obesity in older adults is controversial. Weight loss without exercise could worsen frailty by accelerating the usual age-related decline in muscle and bone mass that leads to sarcopenia and osteopenia, respectively. Because of the important problem of frailty in obese older adults, it is important to determine the most efficacious approach in reducing, or even reversing frailty in this population. The primary objective of this proposal is to evaluate which distinct type of physical exercise (resistance, aerobic, or combined resistance + aerobic) is most efficacious in preventing the weight-loss-induced reduction in muscle and bone mass and reversing frailty in obese older adults.

ELIGIBILITY:
Inclusion Criteria:

* 65-85 years old
* Obese men and women (BMI > or equal to 30 kg/m2)
* Stable weight (±2 kg) during the last 6 mos.
* Must be sedentary (regular exercise <1 h/wk or <2 x/wk for the last 6 mos.)
* Be judged, during the initial screening, to be well motivated and reliable

Exclusion Criteria:

* Any major chronic diseases
* Any condition or unstable diseases that would interfere with exercise or dietary restriction, in which exercise or dietary restriction are contraindicated, or that would interfere with interpretation of results that include but are not limited to:
* Cardiopulmonary disease (e.g., recent MI, unstable angina, stroke etc.)
* Severe orthopedic/musculoskeletal or neuromuscular impairments that would contraindicate participation in exercise
* Visual or hearing impairments that interfere with following directions
* Diagnosis of dementia
* History of malignancy during the past 5 yr
* Recent use of bone acting drugs (e.g. use of estrogen, or androgen containing compound, raloxifene, calcitonin, parathyroid hormone during the past year or biphosphonates during the last two years)
* Individuals on insulin or with a fasting blood glucose of > 140mg/dl, and/or a 2 hour post-glucose of >250 mg/dl
* BMD t-scores of <-2.3 of the lumbar spine and proximal femur
* serum creatinine >2.0 mg/dl
* No commitments, life situations or conditions that would interfere with their participation in the study

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2010-02; Primary Completion 2016-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Physical Function | 6 Months
  The Physical Performance Test includes seven standardized tasks (walking 15.2 m [50 ft], putting on and removing a coat, picking up a penny, standing up from a chair, lifting a book, climbing one flight of stairs, and performing a progressive Romberg test) plus two additional tasks (going up and down four flights of stairs and making a 360-degree turn). The score for each task ranges from 0 to 4, with higher scores indicating better physical performance; a perfect score would be 36.

SECONDARY OUTCOMES:
Change in lean mass | 6 months
  Assessed using dual energy x-ray absorptiometry (DXA)
Change in fat mass | 6 months
  Assessed using DXA
Change in muscle strength | 6 months
  Assessed using 1-repetition maximum and dynamometry
Change in gait speed | 6 months
  Measured as time to walk a certain distance
Change in areal bone mineral density | 6 months
  Assessed by using DXA
Change in biochemical marker for bone turnover and bone metabolism | 6 months
  Assessed by using enzyme linked immunoabsorbent assay and radioimmunoassay
Change in circulating cytokines | 6 months
  Assessed by using enzyme linked immunoassay
Change in adipocytokines | 6 months
  Assessed by using enzyme linked immunoassay
Change in aerobic capacity | 6 months
  Assessed by using indirect calorimetry during graded exercise stress test
Change in systolic and diastolic blood pressure | 6 months
  Assessed by using sphygmomanometer
Change in serum glucose | 6 months
  Assessed by glucose oxidase method
Change in serum lipids | 6 months
  Assessed by automated enzymatic/colorimetric assays
Change in habitual physical activity assessed by questionnaires | 6 months
  Using the Stanford physical activity questionnaire (score range: 0 to 40 with higher scores indicating higher physical activity levels)
Change in habitual physical activity measured objectively | 6 months
  Using accelerometers
Change in serum insulin | 6 months
  Assessed by immunoassay
Change in serum estradiol | 6 months
  Assessed by immunoassay
Change in 25 hydroxyvitamin D | 6 months
  Assessed by immunoassay
Change in Impact of Weight on Quality of Life_Lite (IWQOL-lite) score | 6 months
  Assessed by IWQO-liteL questionnaire
Change in Medical Outcomes 36-Item short form Health survey (SF-36) | 6 months
  Assessed by Physical component summary and mental component summary score (score range 0 to 100, with higher scores indicating better health status)
Change in gene expression of muscle anabolic and catabolic factors | 6 months
  Assessed by reverse transcription polymerase chain reaction and nanostring
Change in protein expression of muscle anabolic and catabolic factors | 6 months
  Assessed by western blotting
Change in concentration of targeted metabolites | 6 months
  Assessed by liquid chromatography hyphenated with mass spectrometry techniques
Change in dynamic balance | 6 months
  Assessed by the obstacle course
Change in static balance | 6 months
  Assessed by one leg stance
Change in modified mini-mental exam | 6 months
  Assessed by using cognitive instrument testing
Change in word fluency | 6 months
  Assessed by using cognitive instrument testing
Change in trail a and trail b | 6 months
  Assessed by using cognitive instrument testing
Change in Ray Auditory verbal learning test | 6 months
  Assessed by using cognitive instrument testing
Change in muscle protein synthesis rate | 6 months
  Assessed by stable isotope methodology
Change in thigh muscle and fat mass | 6 months
  Assessed by magnetic resonance imaging (MRI)
Change in visceral fat mass | 6 months
  Assessed by MRI
Change in mood | 6 months
  Assessed by geriatric depression scale (score range: 0 to 30, where lower scores indicating better mood)
Change in waist circumference | 6 months
  Using a tape measure
Change in serum testosterone | 6 months
  Assessed by immunoassay
Change in subjective ability to function | 6 months
  Assessed by Functional Status Questionnaire (score range: 0 to 36 with higher scores indicating better function)
Change is serum sclerostin | 6 months
  Assessed by immunoassay
Change in parathyroid hormone | 6 months
  Assessed by immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD FACP FACE, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - New Mexico VA Medical Center and University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Colleluori G, Viola V, Bathina S, Armamento-Villareal R, Qualls C, Giordano A, Villareal DT. Effect of aerobic or resistance exercise, or both on insulin secretion, ciliary neurotrophic factor, and insulin-like growth factor-1 in dieting older adults with obesity. Clin Nutr. 2025 Aug;51:50-62. doi: 10.1016/j.clnu.2025.05.016. Epub 2025 May 28. PMID 40527119
- [Derived] Armamento-Villareal R, Aguirre L, Waters DL, Napoli N, Qualls C, Villareal DT. Effect of Aerobic or Resistance Exercise, or Both, on Bone Mineral Density and Bone Metabolism in Obese Older Adults While Dieting: A Randomized Controlled Trial. J Bone Miner Res. 2020 Mar;35(3):430-439. doi: 10.1002/jbmr.3905. Epub 2019 Dec 4. PMID 31797417
- [Derived] Colleluori G, Aguirre L, Phadnis U, Fowler K, Armamento-Villareal R, Sun Z, Brunetti L, Hyoung Park J, Kaipparettu BA, Putluri N, Auetumrongsawat V, Yarasheski K, Qualls C, Villareal DT. Aerobic Plus Resistance Exercise in Obese Older Adults Improves Muscle Protein Synthesis and Preserves Myocellular Quality Despite Weight Loss. Cell Metab. 2019 Aug 6;30(2):261-273.e6. doi: 10.1016/j.cmet.2019.06.008. Epub 2019 Jul 3. PMID 31279675
- [Derived] Villareal DT, Aguirre L, Gurney AB, Waters DL, Sinacore DR, Colombo E, Armamento-Villareal R, Qualls C. Aerobic or Resistance Exercise, or Both, in Dieting Obese Older Adults. N Engl J Med. 2017 May 18;376(20):1943-1955. doi: 10.1056/NEJMoa1616338. PMID 28514618